CLINICAL TRIAL: NCT06718049
Title: Role of Interleukin 18 (IL-18) and Interleukin 18 Binding Protein (IL-18BP) in the Diagnostic Work-up of Systemic Juvenile Idiopathic Arthritis and Autoinflammatory Diseases: Possible Biomarkers in the Differential Diagnosis of Other Febrile Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: REUMAIL18/2020
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Systemic Juvenile Idiopathic Arthritis (sJIA)
Keywords: Systemic Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample for haematochemical analysis and assay of IL-18 and IL-18BP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Literature data suggest that elevated blood values of IL-18 and IL-18 Binding Protein and alterations in their ratio may be significantly correlated with various autoinflammatory diseases, such as systemic juvenile idiopathic arthritis, recurrent autoinflammatory fevers etc. In this view, the clinical implication of this observational, prospective, single-centre, non-pharmacological study will be the definition of new laboratory markers that may be useful in the early differential diagnosis of certain rare and serious paediatric diseases.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the role of IL-18 and IL-18 Binding Protein as biomarkers of systemic Juvenile Idiopathic Arthritis and recurrent autoinflammatory fevers, while the secondary one is to investigate the superiority of IL-18 and IL-18 Binding Protein over other cytokines and inflammatory indexes in the differential diagnosis of systemic Juvenile Idiopathic Arthritis and recurrent fevers of an autoinflammatory nature.

The study will enroll patients referred to the Pediatric Rheumatology Outpatient Clinic of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy, for suspected Juvenile Idiopathic Arthritis or suspected recurrent fever/self-inflammatory disease.

Patients will be enrolled during the acute phase of the disease and, prior to the start of immunosuppressive therapy (i.e. corticosteroids, colchicine, biological drugs), a blood sample will be taken for haematochemical investigations, according to clinical practice, as well as an additional blood sample for the assay of IL-18 and IL-18 Binding Protein.

The following variables will be considered for each patient: demographic data; key clinical features; haemochromocytometric test; liver and kidney function tests; indexes of inflammation and acute phase proteins; inflammatory cytokines panel; serum values of IL-18 and IL-18 Binding Protein.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 years and 18 years;
* Being affected by 1 of the following: Juvenile Idiopathic Arthritis; recurrent fever/ autoinflammatory disease; rheumatic disease; severe infectious diseases (sepsis, meningitis, urinary tract infection, lower respiratory tract infection);
* Obtaining informed consent from parents/legal guardians of paediatric patients.

Exclusion Criteria:

• Patients in whom the suspicion of rheumatic disease is based on a finding of subclinical carditis or chorea.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study enrolls patients referred to the Pediatric Rheumatology Outpatient Clinic of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria of Bologna, Italy, for suspected Juvenile Idiopathic Arthritis or suspected recurrent fever/self-inflammatory disease.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum levels of IL-18, and IL-18BP | at T0 - T1(3 months) - T2(12 months)
  pg/mL

SECONDARY OUTCOMES:
Serum levels of inflammatory cytokines | at T0 - T1(3 months) - T2(12 months)
  IL-6; IL-8; TNF alpha; IL-12p70; IL-1 beta; IL-10 (pg/mL)
Serum levels of acute phase proteins | at T0 - T1(3 months) - T2(12 months)
  C-reactive protein (mg/dL); amyloid A protein (mg/dL); ferritin (ng/dL); transferrin (mg/dL); fibrinogen (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Miniaci, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy